CLINICAL TRIAL: NCT05387668
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of BGB-23339 in Healthy Japanese and Caucasian Subjects
Brief Title: Safety, Tolerability, and Pharmacokinetics of BGB-23339 in Healthy Japanese and Caucasian Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor determined the data was no longer needed.
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: BGB-23339-102
Record Dates: First submitted 2022-05-18; First posted 2022-05-24 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Japanese cohort (Experimental): Three ascending dose levels of either BGB-23339 or placebo.
  Interventions: Drug: BGB-23339; Drug: Placebo
- Part B: Caucasian cohort (Experimental): One dose level of either BGB-23339 or placebo based on data collected in Part A.
  Interventions: Drug: BGB-23339; Drug: Placebo

INTERVENTIONS:
Drug: BGB-23339 — Administered orally as a tablet.
Drug: Placebo — Administered orally as a tablet.

SUMMARY:
This study is designed to evaluate the influence of ethnic factors on the safety, tolerability, and pharmacokinetics (PK) of BGB-23339 after multiple dosing under fasting condition in healthy Japanese and Caucasian participants.

DETAILED DESCRIPTION:
The study comprises 2 parts: Part A is a randomized, double-blind, placebo-controlled, multiple ascending dose study to evaluate the safety, tolerability, and PK profile of BGB-23339 in healthy Japanese subjects. Part B is a randomized, double-blind, placebo-controlled, multiple-dose study to evaluate the safety, tolerability, and PK profile of BGB-23339 in healthy Caucasian subjects.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all of the following inclusion criteria to be considered eligible for participation in this study:

1. Signed informed consent form (ICF) and able to comply with study requirements
2. Healthy Japanese or Caucasian men and/or women of no childbearing potential aged ≥ 18 years and ≤ 55 years on the day of signing the ICF (or the legal age of consent), and to be specific:

   1. For Part A only: Eligible Japanese subjects should have both biological parents and 4 biological grandparents of Japanese descent, and their 4 biological grandparents must be born in Japan.
   2. For Part B only: Eligible Caucasian subjects should 1) have both biological parents and 4 biological grandparents of Caucasian descent, and 2) be matched by body weight (± 20% body weight [kg]), height (± 15% height [centimeter (cm)]) and sex to each Japanese subject receiving the highest dose level planned in Part A.
3. Subjects are in good general health as determined by the investigator or medically qualified designee, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from this study:

Medical Conditions

1. History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study drug; or interfering with the interpretation of data
2. Active herpes infection, including herpes simplex 1 and 2 and herpes zoster (demonstrated on physical examination and/or medical history ≤ 2 months before randomization)
3. Any malignancies within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
4. Positive HBV, HCV and HIV test
5. History or risk for tuberculosis (TB)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-10-17 (Estimated); Study Completion 2022-10-17 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Duration of Study (Up to 11 weeks)
  Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), including laboratory values, vital signs, and electrocardiogram results.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) of BGB-23339 from time zero to last quantifiable time (AUClast) quantifiable time (AUClast) | Up to Day 10
Area under the plasma concentration-time curve (AUC) of BGB-23339 from time zero to end of dosing interval (AUCtau) | Up to Day 10
Maximum observed plasma concentration (Cmax) of BGB-23339 | Up to Day 10
Time to maximum plasma concentration (Tmax) of BGB-23339 | Up to Day 10
Trough plasma concentration (Ctrough) of BGB-23339 | Up to Day 10
Apparent terminal elimination half-life (t½) of BGB-23339 | Up to Day 10
Apparent systemic clearance (CL/F) of BGB-23339 | Up to Day 10
Apparent volume of distribution (Vz/F) of BGB-23339 | Up to Day 10
Metabolite to parent ratio for BGB-23339 and its metabolite BGB-25808 | Up to Day 10

CONTACTS AND LOCATIONS:
Locations (1):
- PPD, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Undecided